CLINICAL TRIAL: NCT02308072
Title: A Phase I Trial of Olaparib in Addition to Cisplatin-based Concurrent Chemoradiotherapy for Patients With High Risk Locally Advanced Squamous Cell Carcinoma of the Head and Neck (NHSCC)
Brief Title: Phase I Study of Olaparib Combined With Cisplatin-based Chemoradiotherapy to Treat Locally Advanced Head and Neck Cancer
Acronym: ORCA-2
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Cancer Research UK (Other); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCL/13/0696; 2014-002525-35 (EudraCT Number)
Record Dates: First submitted 2014-12-02; First posted 2014-12-04 (Estimated); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Head and Neck Cancer
Keywords: Squamous Cell Carcinoma; Head and Neck Cancer; Locally Advanced; Olaparib; Cisplatin; IMRT; Chemoradiotherapy; PARP; HNSCC
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell; Squamous Cell Carcinoma of Head and Neck | interventions — olaparib; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Olaparib + Cisplatin + IMRT (Experimental): Olaparib: 50, 100, 150 or 200 mg twice a day for between 3-5 sequential days, depending on cohort allocation, in combination with Cisplatin: 35 mg/m^2 on day 1, and IMRT: 2 Gy radiotherapy given on days 1-5
  Treatment will start on day 1 of every week. Patients will receive up to 7 weeks of combination chemotherapy and radiotherapy treatment.
  Interventions: Drug: Olaparib; Drug: Cisplatin; Radiation: IMRT

INTERVENTIONS:
Drug: Olaparib — 50 mg, 100 mg, 150 mg or 200 mg taken twice daily (depending on dose under investigation at time of registration) on days 1-3, 1-4 or 1-5 (depending on allocation of treatment schedule) of each week of treatment.
Drug: Cisplatin — 35 mg/m^2 IV on day 1 of each week of treatment during radiotherapy for a total of 7 weeks (total overall dose 245 mg/m^2)
Radiation: IMRT — 2 Gy delivered in 35 fractions, on days 1-3, 1-4 or 1-5 each week for up to 7 weeks (total overall dose delivered 70 Gy)

SUMMARY:
The phase I trial aims to determine the recommended phase II dose (RP2D) and schedule of olaparib in combination with standard cisplatin-based chemoradiotherapy, in patients with high-risk locally advanced squamous cell carcinoma of the head and neck (HNSCC), by assessing the safety and tolerability of the treatment combination.

DETAILED DESCRIPTION:
ORCA-2 is a phase I trial in patients with locally advanced, with or without metastatic nodal disease.

Patients will receive olaparib (a PARP inhibitor) in combination with standard cisplatin-based chemotherapy and intensity modulated radiotherapy (IMRT).

Olaparib, cisplatin and radiotherapy will be given in combination every week for a maximum of 7 weeks. Prior to starting combination treatment, olaparib will be started 7 days before the first week of combination treatment. Olaparib will be given twice daily on days 1-3 of each week of treatment (either alone during week 0 or in combination with chemotherapy and radiotherapy during weeks 1-7). Cisplatin will be started on day 1 of each week, and given once a week during radiotherapy treatment for a total of 7 weeks. Radiotherapy will be delivered on days 1-5 of each week using IMRT, for a total of 7 weeks.

The phase I trial aims to determine the recommended phase II dose of olaparib (50mg, 100mg, 150mg or 200mg bd) - the dose of olaparib patients receive will depend on the dose under investigation at the time of patient registration.

Dose escalation will be guided by the two-dimensional dose escalation design called Product of Independent Beta Probabilities escalation (PIPE). It will recommend the choice of dose/duration combination cohort of olaparib for subsequent patients by estimating the contour that divides dose/duration combination cohorts to be those above the target toxicity rate (equal to 33%) and those below. The recommended phase II cohort(s) are those that have been experimented on during the trial and are also closest to (but not above) the estimated contour calculated using all trial data.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed high-risk locally advanced HNSCC, patients who would normally be offered cisplatin-based radical chemoradiotherapy
2. Estimated life expectancy of at least 16 weeks
3. WHO performance status 0 or 1
4. Aged ≥18 years
5. Adequate bone marrow function: absolute neutrophils grade 0 or 1, platelets grade 0 or 1, haemoglobin grade 0 or 1
6. Adequate renal function: Creatinine grade 0 or 1, Calculated GFR ≥60 mL/min (if calculated value is <60 mL/min then an isotope GFR assessment should be performed or an estimation from 24h urine collection)
7. Adequate liver function: Serum bilirubin grade 0 or 1, AST or ALT grade 0 or 1
8. Patients must be able to swallow olaparib tablets
9. Willing to use contraception for the duration of the trial treatment and for six months after completion of treatment
10. Able to give informed consent
11. Patients willing and able to comply with the protocol for the duration of the study

Exclusion Criteria:

1. Head & neck cancers of the following types: Nasopharyngeal and paranasal sinus tumours, Oral squamous cell carcinomas (tumours of the oral cavity), Low risk Human Papilloma Virus positive oropharyngeal tumours (tonsillar and tongue base tumours)
2. Confirmed distant metastatic disease
3. Previous chemotherapy or radiotherapy for the treatment of HNSCC tumour
4. Previous therapy with a PARP inhibitor
5. Chemotherapy, immunotherapy or radiotherapy within 28 days prior to registration
6. Prior history of malignancy, except for basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, breast or prostate. Patient must have been free of malignancy for a period of 3 years prior to first dose of trial drug
7. Women who are pregnant or lactating
8. Pre-existing gastrointestinal disorders that may interfere with the delivery or absorption of olaparib
9. Grade 3 or 4 peripheral neuropathy - If considered significant by the treating clinician a lower grade neuropathy may be considered as exclusion criterion
10. Significant hearing difficulties or tinnitus (deaf patients can be included) - Whilst not excluded, patients with mildly impaired hearing or tinnitus must be made aware of potential ototoxicity and may choose not to be included. If included, it is recommended that audiograms be carried out at baseline.
11. Any serious and/or unstable pre-existing medical, psychiatric or other condition that, in the treating clinician's judgment, could interfere with patient safety or obtaining informed consent
12. Known hepatitis B or C infection (testing for Hepatitis and HIV for the trial is not mandatory)
13. Immunocompromised patients (e.g. known HIV positive status)
14. Active uncontrolled infection
15. The current use of drugs which are known to inhibit or induce CYP3A4
16. Resting ECG with QTc > 470msec on 2 or more time points within a 24 hour period or family history of long QT syndrome.
17. Patients with myelodysplastic syndrome/acute myeloid leukaemia.
18. Patients with a known hypersensitivity to olaparib or any of the excipients of the product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Dose Limiting Toxicity | From start of week 1 to 6 weeks after end of combination treatment (combination treatment = 7 weeks)
  Detailed adverse event monitoring will be conducted according to CTCAE v4.03. Dose Limiting Toxicity (DLT) is defined as any adverse event or laboratory abnormality detailed in the trial protocol, that is considered to be trial treatment related and commencing anytime during the DLT evaluation period (from start of week 1 of olaparib + CRT until 6 weeks after end of olaparib + CRT).

SECONDARY OUTCOMES:
Occurrence and Severity of Adverse Events | From date of registration until 12 weeks after completion of trial treatment
  Will include all grade 1-5 adverse events
Best Overall Response | Determined from imaging/scans performed pre-registration, during treatment and follow-up until disease progression or up to 2 years from date of registration
  Response will be assessed according to RECIST v1.1. Confirmation of complete or partial response is not required.
Time to Loco-Regional Progression | From date of registration to date of documented disease progression, assessed up to 2 years from date of registration
  Time to loco-regional progression will be evaluated from the date of trial entry to date of documented disease progression according to RECIST v1.1 or histological/cytological confirmation.
Time to Progression | From date of registration to date of documented objective disease progression
  Time to progression will be determined from the date of patient registration to objective disease progression according to RECIST v1.1
Progression Free Survival | From date of registration to date of documented disease progression or death from any cause, whichever comes first. Assessed up to 2 years from date of registration.
  Progression-free survival will be calculated from the date of trial entry to the date of documented disease progression, or death from any cause. Where progression is suspected and subsequently confirmed by scans, the date of documented suspected progression will be used.
Overall Survival | From date of registration until date of death or date of last follow-up assessment (up to 2 years from date of registration)
  Overall survival time will be calculated from the date of trial entry to the date of death from any cause or end of trial follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Forster, Principal Investigator — University College, London
Locations (3):
- United Kingdom (3):
  - Guy's and St Thomas' NHS Foundation Trust, London
  - University College London Hospitals NHS Foundation Trust, London
  - Velindre Cancer Centre, Wales

IPD SHARING:
Plan to Share IPD: Undecided